CLINICAL TRIAL: NCT00129428
Title: The Effectiveness of UVB Irradiation in the Treatment of Skin Conditions With Altered Dermal Matrix: An Open Pilot Study
Brief Title: Ultraviolet B (UVB) Light Therapy in the Treatment of Skin Conditions With Altered Dermal Matrix
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Clinical Lecturer in Dermatology, Medical School Department, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Derm 447
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Keloid; Scleroderma, Localized; Acne Keloidalis; Scars; Granuloma Annulare
Keywords: UVB; keloid; scleroderma; acne keloidalis nuchae; scars; granuloma annulare
MeSH Terms: conditions — Keloid; Scleroderma, Localized; Acne Keloid; Cicatrix; Granuloma Annulare; Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UVB Irradiation (Experimental): A dose of up to 320 mJ/cm2 from a UVB irradiation device will be administered at maximum 5 times per week for 16 weeks.
  Interventions: Procedure: UVB Irradiation

INTERVENTIONS:
Procedure: UVB Irradiation — A dose of up to 320 mJ/cm2 from a UVB irradiation device will be administered at maximum 5 times per week for 16 weeks.

SUMMARY:
This research study will evaluate the effectiveness of high dose UVB light therapy in the treatment of keloid (or hypertrophic scar), scleroderma, acne keloidalis nuchae, old burn scars, granuloma annulare or related conditions.

DETAILED DESCRIPTION:
Keloid, scleroderma, acne keloidalis nuchae, and burn scars are all characterized by collagenous thickening of the skin resulting in superficial and deep cutaneous sclerosis. Treatments for these disabling conditions are inadequate at present. Recently, in non-controlled studies, UVA1 was shown to induce improvement in patients with scleroderma, granuloma annulare and urticaria pigmentosa.

However, UVA1 is unable to penetrate pigmented skin at an effective level to activate matrix metalloproteinases (MMPs). The investigators' preliminary data show that high dose UVB (160 mJ/cm2) will penetrate pigmented skin and activate the cellular pathways necessary to stimulate MMPs. They postulate, therefore, that in pigmented skin, higher than usual UVB doses can improve these fibrosing skin conditions safely through collagenase-mediated removal of excess dermal collagen via activation of MMP pathways.

The purpose of this research project is to study the effectiveness of high dose UVB (290-320nm at up to 320mJ/cm2) irradiation for the treatment of skin conditions with altered dermal matrix in patients with increased skin pigmentation. These disorders include but are not limited to keloid (or hypertrophic scar), scleroderma, acne keloidalis nuchae, old burn scars, and granuloma annulare. Up to fifty patients with one of these diagnoses or related conditions will receive UVB irradiation up to 5 times per week, for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* In good general health and between 10-80 years of age.
* Willing and able to receive UVB, as directed in the protocol; make evaluation visits; follow protocol restrictions; and sign a written, witnessed, informed consent form.
* Have a clinical diagnosis of keloid, scleroderma, old burn scars, granuloma annulare, or acne keloidalis nuchae.
* No disease states or physical conditions that would impair evaluation of the test site
* Must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* Have a history of photosensitivity (development of hives or bumps with exposure to light) or experience hypersensitivity in a UVB photo-provocation test.
* Have participated in another investigational study in the past 4 weeks, taken oral therapy for skin condition, or on photosensitizing medications.
* Pregnant, nursing, or planning to become pregnant during the study.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Improvement in appearance of keloids (hypertrophic scars), scleroderma, acne keloidalis nuchae,old burn scars, granuloma annulare, and related conditions with altered dermal matrix | Subjects will be evaluated at weeks 1, 2, 4, and then at monthly intervals until the end of the study.

SECONDARY OUTCOMES:
Assays to be performed on biopsy specimens may include any or all of the following assays: in situ hybridization, immunohistologic analysis, in situ zymography, radioimmunoassay, and Western blot analysis | Assays will be performed after specimen collection
Photographs will also be taken. | At baseline and at end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States